CLINICAL TRIAL: NCT04461002
Title: Evaluation of the Correlation Between Molecular Phenotype and Radiological Signature (by PET-scanner and MRI) of WHO II and III Grade Incident Gliomas.
Brief Title: Evaluation of the Correlation Between Molecular Phenotype and Radiological Signature (by PET-scanner and MRI) of Incident WHO II and III Grade Gliomas.
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: RadioGLioSign
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Retrospective cohort
  Interventions: Other: Retrospective analysis

INTERVENTIONS:
Other: Retrospective analysis — Evaluate the correlation between tumour molecular profile and preoperative imaging data (FDG and FDOPA PET-scan and multimodal MRI).

SUMMARY:
From the medical records of a series of patients operated on for incident grade II and III glioma, the primary objective is to evaluate the correlation between the molecular profile of tumours and preoperative imaging data (by FDG and FDOPA PET-scan and multimodal MRI).

DETAILED DESCRIPTION:
A retrospective monocentre study of medical data (clinical, histological, molecular and imaging) contained in the medical records of patients operated on for Grade II or III incident glioma.

ELIGIBILITY:
Inclusion Criteria:

* Subject 18 years of age or older, having been informed of the research
* Subject operated on with an incident glioma of grade II or III, histologically confirmed (WHO 2016 classification)
* Subject for which all preoperative imaging data is available (MRI, FDG and FDOPA PET-scan)
* Subject for which molecular data of the lesion are available

Exclusion Criteria:

* Subject having signified his opposition to the use of his medical data
* Subject under safeguard of justice, guardianship or trusteeship
* Subject with incomplete or missing part of the molecular and/or imaging data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population represents the totality of patients with a glioma surgery in the centre between February 2015 and May 2019, with a complete and usable medical file.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Primary outcome | 4 years
  Evaluate the correlation between tumour molecular profile and preoperative imaging data (FDG and FDOPA PET-scan and multimodal MRI).

SECONDARY OUTCOMES:
Molecular profile | 4years
  Evaluate the overall survival and progression-free survival of patients based on the molecular profile of gliomas.
Imaging data | 4 years
  To evaluate the overall survival and progression-free survival of patients based on imaging data (PET-scan and MRI) of gliomas.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe METELLUS, MD PD, Principal Investigator — Hôpital Privé Clairval
Locations (1):
- Hôpital Privé Clairval, Marseille, France

IPD SHARING:
Plan to Share IPD: No